CLINICAL TRIAL: NCT03366181
Title: SGLT2i As Anti Arrhythmic Therapies and Sudden Cardiac Death in Implantable Cardioverter Defibrillators (ICDs) Recipients
Brief Title: SGLT2i As Anti Arrhythmic Therapy to Prevent Sudden Cardiac Deaths.
Status: Completed | Type: Observational
Sponsor: University of Campania Luigi Vanvitelli (Other)
Responsible Party: Principal Investigator, Celestino Sardu, Associate Professor, University of Naples
Other Study IDs: 10.12.2017.2
Record Dates: First submitted 2017-11-28; First posted 2017-12-08 (Actual); Last update posted 2025-01-20 (Actual); Status verified 2025-01

CONDITIONS: Heart Failure; ICD; Diabetes Mellitus Type 2; SGLT2i
MeSH Terms: conditions — Heart Failure; Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Heart failure patients with T2DM and treated with ICD under SGLT2i therapy.: These patients with T2DM and stable heart failure were previously treated with ICD, and received a SGLT2i therapy. These patients were named SGLT2i-users.
- Heart failure patients with T2DM and treated with ICD and without SGLT2i therapy.: Heart failure patients with T2DM and treated with ICD that did not receive the SGLT2i therapy. These patients were named Non-SGLT2i users.

SUMMARY:
Failing heart negative remodeling alterations might provide electrical heterogeneity and cardiac remodeling, thus potentially contributing to the occurrence of ventricular arrhythmia and subsequent sudden cardiac death (SCD). In this study we have prospectively investigated whether sodium glucose transporte-2 inhibitors (SGLT2i) could modulate serum markers of heart failure (ultra sensitive Troponin , B type Natriuretic Peptide (BNP), C reactive protein (CRP), the heart rate (HR) and serum catecholamines in patients with type 2 diabetes mellitus (T2DM), and be used as predictors for the occurrence of malignant ventricular arrhythmias (VTAs) in patients who had received an Implantable Cardioverter Defibrillator (ICD) for primary prevention. In these T2DM patients with ICD we investigated the functionality of devices, the appropriate and inappropriate shocks, and the hospitalizations for heart failure and the cardiac deaths.

ELIGIBILITY:
Inclusion Criteria:

* stable heart failure; indication for a ICD and/or a CRT-d system; NYHA Class II-III; left ventricle ejection fraction <35%; patients receiving optimal medical therapy without controindications to receive SGLT2i; diagnosis of T2DM.

Exclusion Criteria:

* NYHA Class I, and IV; co-morbidities which may limit life to <6 months; history of cardiac surgery or intervention within the preceding 90 days; history of moderate to severe chronic obstructive pulmonary disease (COPD), defined as needing chronic oxygen therapy, or recent (within 30 days) hospitalization for COPD flare-up; pregnancy; history of primary pulmonary hypertension.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: heart failure patients with reduced LVEF (LVEF <35%) and affected by T2DM, previously treated with ICD and indication to receive SGLT2i therapy.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2017-11-20 (Actual); Study Completion 2017-11-26 (Actual)

PRIMARY OUTCOMES:
cardiac deaths | 12 months
  authors will report cardiac deaths by hospital discarge schedules, visits, telephonic interviews, and deaths registry.
Heart failure hospitalization | 12 months
  authors will report heart failure hospitalization by hospital discarge schedules, visits, telephonic interviews.
ICDs' intervention | 12 months
  authors will report ICDs' intervention by hospital discarge schedules, visits, telephonic interviews, and telemetric devices interrogations.

SECONDARY OUTCOMES:
arrhythmic burden | 12 months
  authors will report arrhythmic burden by hospital discarge schedules, visits, telephonic interviews, egg hollering, and telemetric devices interrogations.

CONTACTS AND LOCATIONS:
Locations (1):
- Raffaele Marfella, Naples, Italy, Italy

IPD SHARING:
Plan to Share IPD: Undecided